CLINICAL TRIAL: NCT00005142
Title: Etiology and Prevalence of Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1013; R01HL022255 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases; Arterial Occlusive Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases; Arterial Occlusive Diseases

SUMMARY:
To determine the prevalence of peripheral arterial disease in a defined population by non-invasive techniques; to evaluate the association of cardiovascular disease risk factors with peripheral vascular disease; to determine whether non-invasive tests of peripheral arterial disease can be utilized as markers for coronary heart disease; to determine the status of the microvasculature using conjunctival photographs and to compare the results with risk factors and the peripheral arterial disease testing results.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerosis is frequently generalized, affecting blood vessels in various parts of the body. Previous studies had noted the strong association between peripheral arterial disease and coronary heart disease and the similarity of risk factors, particularly diabetes and cigarette smoking for both diseases. The natural history of peripheral arterial disease had not been delineated because of the lack, until recently, of accurate and reliable non-invasive testing.

DESIGN NARRATIVE:

All 624 subjects were initially studied under a Lipid Research Clinic protocol that involved two evaluations, visit 1 and visit 2. At visit 2, half of the subjects were from a random sample of the LRC visit 1 cohort and others were selected from the visit 1 cohort for hyperlipidemia, defined as being at or above age- and sex-specific 90th percentiles for cholesterol or 95th percentiles for triglycerides or taking lipid-lowering medications. At visit 2, the subjects were characterized as to age; sex; drug, diet, alcohol and smoking history; personal and family history of cardiovascular disease; Rose questionnaire; and electrocardiogram and examination by a cardiologist. The subjects were given a traditional manual examination for peripheral arterial disease and four non-invasive tests including segmental blood pressure, flow velocity by Doppler ultrasound, postocclusive reactive hyperemia, and pulse reappearance half-time. The subjects were categorized into large vessel peripheral arterial disease, isolated small vessel peripheral arterial disease or normal based on the results of non-invasive testing and followed for an average of four years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1978-07; Study Completion 1990-03 (Actual)

REFERENCES:
- [Background] Criqui MH, Fronek A, Barrett-Connor E, Klauber MR, Gabriel S, Goodman D. The prevalence of peripheral arterial disease in a defined population. Circulation. 1985 Mar;71(3):510-5. doi: 10.1161/01.cir.71.3.510. PMID 3156006
- [Background] Criqui MH, Fronek A, Klauber MR, Barrett-Connor E, Gabriel S. The sensitivity, specificity, and predictive value of traditional clinical evaluation of peripheral arterial disease: results from noninvasive testing in a defined population. Circulation. 1985 Mar;71(3):516-22. doi: 10.1161/01.cir.71.3.516. PMID 3156007
- [Background] Baker LL, Criqui MH. High- and low-density lipoprotein cholesterol: correlates in an older population. Prev Med. 1985 Mar;14(2):155-64. doi: 10.1016/0091-7435(85)90030-1. PMID 4048078
- [Background] Criqui MH, Coughlin SS, Fronek A. Noninvasively diagnosed peripheral arterial disease as a predictor of mortality: results from a prospective study. Circulation. 1985 Oct;72(4):768-73. doi: 10.1161/01.cir.72.4.768. PMID 4028377
- [Background] Standeven M, Criqui MH, Klauber MR, Gabriel S, Barrett-Connor E. Correlates of change in postmenopausal estrogen use in a population-based study. Am J Epidemiol. 1986 Aug;124(2):268-74. doi: 10.1093/oxfordjournals.aje.a114385. PMID 3728443
- [Background] Barrett-Connor E, Criqui MH, Witztum JL, Philippi T, Zettner A. Population-based study of glycosylated hemoglobin, lipids, and lipoproteins in nondiabetic adults. Arteriosclerosis. 1987 Jan-Feb;7(1):66-70. doi: 10.1161/01.atv.7.1.66. PMID 3813976
- [Background] Criqui MH, Lee ER, Hamburger RN, Klauber MR, Coughlin SS. IgE and cardiovascular disease. Results from a population-based study. Am J Med. 1987 May;82(5):964-8. doi: 10.1016/0002-9343(87)90159-8. PMID 3578366
- [Background] Criqui MH, Browner D, Fronek A, Klauber MR, Coughlin SS, Barrett-Connor E, Gabriel S. Peripheral arterial disease in large vessels is epidemiologically distinct from small vessel disease. An analysis of risk factors. Am J Epidemiol. 1989 Jun;129(6):1110-9. doi: 10.1093/oxfordjournals.aje.a115233. PMID 2786328
- [Background] Criqui MH, Langer RD, Fronek A, Feigelson HS. Coronary disease and stroke in patients with large-vessel peripheral arterial disease. Drugs. 1991;42 Suppl 5:16-21. doi: 10.2165/00003495-199100425-00005. PMID 1726213
- [Background] Criqui MH, Langer RD, Fronek A, Feigelson HS, Klauber MR, McCann TJ, Browner D. Mortality over a period of 10 years in patients with peripheral arterial disease. N Engl J Med. 1992 Feb 6;326(6):381-6. doi: 10.1056/NEJM199202063260605. PMID 1729621